CLINICAL TRIAL: NCT07087405
Title: Stretch Mark Treatment Using Subcutaneous Skin Abrasion
Brief Title: Striae Distensae Treatment Using Deep Skin Abrasion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Arin Greene, Professor of Surgery, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00051021
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Striae Distensae
Keywords: Striae Distensae
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Striae Distensae Treatment (Experimental): Striae Distensae Treatment With A Device
  Interventions: Device: Striae Distensae Treatment Device

INTERVENTIONS:
Device: Striae Distensae Treatment Device — One time deep skin treatment

SUMMARY:
The goal of this clinical trial is to learn if a device works to treat striae distensae. It will also learn about the safety of the device. The main questions it aims to answer are:

1. Does the device improve the appearance of striae distensae?
2. Does the device cause any problems when treating striae distensae? Researchers will compare the appearance of striae distensae before and after treatment with the device.

Participants will:

1. Undergo treatment with the device in the clinic
2. Visit the clinic 1 week, 3 months, and 1 year for checkups and tests

DETAILED DESCRIPTION:
Participants will have the area of striae distensae anesthetized with local anesthetic. A biopsy will be performed and a device will be placed underneath the skin that will abrade the skin. Three months later another biopsy will be performed, photographs will be taken, and participants will fill out surveys to determine the effectiveness of the device to improve the appearance of the striae distensae.

ELIGIBILITY:
Inclusion Criteria:

* Striae distensae

Exclusion Criteria:

* Smoking, coagulation deficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in Striae Distensae Appearance | From enrollment to 12 months after treatment
  Comparison of photographs before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Arin Greene, MD, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: No
IPD will be aggregated